CLINICAL TRIAL: NCT02479893
Title: Cold Snare Polypectomy vs Hot Snare Polypectomy vs APC for the Complete Removal of Left Sided Colon Polyps. A Prospective,Randomized Trial
Brief Title: Cold Snare,Hot Snare and APC Polypectomy for the Complete Removal of Small Left Sided Colon Polyps
Status: Completed | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Collaborators: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Nikos Viazis, Director gastroenterologist, Evangelismos Hospital
Other Study IDs: 80/30-04-2015
Record Dates: First submitted 2015-05-26; First posted 2015-06-24 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Colonic Polyps
Keywords: cold snare polypectomy; APC; hot snare polypectomy
MeSH Terms: conditions — Colonic Polyps | interventions — Sigmoidoscopy; Colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colonic polyps tissue samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- cold snare polypectomy: CSP: In this group polyps will be removed with the cold snare polypectomy technique, as a single piece. Additionally, a 1-2mm of normal tissue around the small polyp will also be ensnared in the CSP.
  Interventions: Procedure: polypectomy
- hot snare polypectomy: HSP: In this group polyps will be removed with the hot snare polypectomy technique as a single piece with a electrosurgical snare and monopolar current with a setting of 30-35 W in the endocut function.
  Interventions: Procedure: polypectomy
- APC polyp destruction-polypectomy: APC: In APC group polyps will be cauterized by application of high power argon plasma coagulation on small waves at 50-60W and flow at 2lt/min,as result the polyp destruction.
  Interventions: Procedure: polypectomy

INTERVENTIONS:
Procedure: polypectomy — Polyps size up to 0.8 cm will removed from the left colon.Re examination in 6 months period with biopsy from the scar of polypectomy.
  Other Names: sigmoidoscopy; colonoscopy

SUMMARY:
Given the limited existing data regarding the advantages and limitations of the existing techniques in the removal of colonic polyps the investigators designed a prospective study in order to compare cold snare vs hot snare vs argon plasma coagulation for the compete removal of colonic polyps of the left colon up to a diameter of 0.8cm.

DETAILED DESCRIPTION:
Adenomatous polyps are the most common neoplastic findings discovered in subjects who undergo colonoscopy either for colorectal screening or during a diagnostic work-up for symptoms.

Currently small polyps 0.3-0.8cm are removed using hot snare polypectomy (HSP) cold snare polypectomy (CSP) while argon plasma coagulation (APC) has been proposed for the cauterization of bigger polyps ("Melt Effect") Endoscopic polypectomy is associated with potential complications, i.e. perforation and bleeding while some polyps may recur after polypectomy.

Given the limited existing data regarding the advantages and limitations of the existing techniques in the removal of colonic polyps the investigators designed a prospective study in order to compare the above mentioned methods for the compete removal of colonic polyps 0,3-0,8 cm from the left side colon.

METHODS The study will be conducted in the endoscopy unit of "Evangelismos" Hospital and in D Surgical clinic of the University Hospital "Attikon".All consecutive patients with colorectal polyps of the left colon (up to the splenic flexure) with a diameter of 0.3-0.8cm will be prospectively randomized to three groups.

1. CSP: In this group polyps will be removed with the cold snare polypectomy technique, as a single piece. Additionally, a 1-2mm of normal tissue around the small polyp will also be ensnared in the CSP.
2. HSP: In this group polyps will be removed with the hot snare polypectomy technique as a single piece with a electrosurgical snare and monopolar current with a setting of 30-35 W in the endocut function.
3. APC: In APC group polyps will be cauterized by application of high power argon plasma coagulation on small waves at 50-60W and flow at 2lt/min.

All polyps will be elevated by submucosal injection of normal saline (1ml) and consequently a special dye (1ml) containing carbon particles (Spot) before applying any of the three removal techniques.

The injection solution protects from thermal injury of deeper layers during the application of current and APC,also the injection of the dye (tattoo) at the polypectomy, ensures that the endoscopist will detect the point of polypectomy in the follow up colonoscopy after 3-6 months.

Spot (GI supply,Camp Hill,PA) is the only commercially available suspension for endoscopic tattooing approved by the Food and Drug Association (FDA). It contains prediluted sterile syrings that are filled with highly purified fine carbon particles ready for endoscopic use.

The study excluded patients with a history of familial polyposis (FAP), Gardner's syndrome, Peutz-Jeghers syndrome, patients with colon Cancer as well as patients with idiopathic inflammatory bowel disease (IBD).

Statistical analysis showed that the sample required to give medium (W = 0.3) the difference between the three groups is 108 patients, with significance level of 5% and validity of the study 80% All patients included in the study will undergo a repeat colonoscopy in a 3-6 month time period. The endoscopist based on tattoos have been received on the first endoscopy during polypectomy will receive multiple biopsies from the point, which will be sent for histological examination.The pathologist will then examine the tissue sample and will define whereas the polyp has been completely eradicated or recurred.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with colorectal polyps of the left colon (up to the splenic flexure) with a diameter of 0.3-0.8cm.

Exclusion Criteria:

* The study excluded patients with a history of familial polyposis (FAP), Gardner's syndrome, Peutz-Jeghers syndrome, patients with colon Cancer as well as patients with idiopathic inflammatory bowel disease (IBD).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with colonic left sided small polyps
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2015-01; Primary Completion 2019-03 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Complete removal of colonic polyps | at 6 months after polypectomy
  The resections margin of the polyp was isolated from the rest of the polyp,stained with black and examined through multiple histological sections in order to certify that no dysplastic cells were traced upon the resection margin.Since all adenoma cases exhibited low grade epithelial dysplasia, as positive margin was considered the presence of dysplastic cell exactly upon the resection margin/black ink.

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Viazis, Director, Principal Investigator — Evangelismos Hospital
Locations (1):
- Evangelismos Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schneider R, Goldman AB, Insall JN. Knee prostheses. Semin Roentgenol. 1986 Jan;21(1):29-46. doi: 10.1016/0037-198x(86)90007-6. No abstract available. PMID 3513321
- [Background] Tolliver KA, Rex DK. Colonoscopic polypectomy. Gastroenterol Clin North Am. 2008 Mar;37(1):229-51, ix. doi: 10.1016/j.gtc.2007.12.009. PMID 18313548
- [Background] Uno Y, Obara K, Zheng P, Miura S, Odagiri A, Sakamoto J, Munakata A. Cold snare excision is a safe method for diminutive colorectal polyps. Tohoku J Exp Med. 1997 Dec;183(4):243-9. doi: 10.1620/tjem.183.243. PMID 9549824
- [Background] Winawer SJ, Zauber AG, Fletcher RH, Stillman JS, O'Brien MJ, Levin B, Smith RA, Lieberman DA, Burt RW, Levin TR, Bond JH, Brooks D, Byers T, Hyman N, Kirk L, Thorson A, Simmang C, Johnson D, Rex DK; US Multi-Society Task Force on Colorectal Cancer; American Cancer Society. Guidelines for colonoscopy surveillance after polypectomy: a consensus update by the US Multi-Society Task Force on Colorectal Cancer and the American Cancer Society. Gastroenterology. 2006 May;130(6):1872-85. doi: 10.1053/j.gastro.2006.03.012. PMID 16697750
- [Background] Metz AJ, Moss A, McLeod D, Tran K, Godfrey C, Chandra A, Bourke MJ. A blinded comparison of the safety and efficacy of hot biopsy forceps electrocauterization and conventional snare polypectomy for diminutive colonic polypectomy in a porcine model. Gastrointest Endosc. 2013 Mar;77(3):484-90. doi: 10.1016/j.gie.2012.09.014. Epub 2012 Nov 27. PMID 23199650
- [Background] Tsiamoulos ZP, Bourikas LA, Saunders BP. Endoscopic mucosal ablation: a new argon plasma coagulation/injection technique to assist complete resection of recurrent, fibrotic colon polyps (with video). Gastrointest Endosc. 2012 Feb;75(2):400-4. doi: 10.1016/j.gie.2011.09.003. Epub 2011 Dec 7. PMID 22154411
- [Background] Anderloni A, Jovani M, Hassan C, Repici A. Advances, problems, and complications of polypectomy. Clin Exp Gastroenterol. 2014 Aug 30;7:285-96. doi: 10.2147/CEG.S43084. eCollection 2014. PMID 25210470
- [Derived] Varytimiadis L, Viazis N, Gkolfakis P, Tribonias G, Tziatzios G, Kyriakopoulos G, Argyrakos T, Pontas C, Papastergiou V, Arkadopoulos N, Smyrniotis V, Mantzaris GJ, Papanikolaou IS. Cold snare polypectomy vs. hot snare polypectomy vs. argon plasma coagulation for small (5-9mm) left-sided colorectal polyps: a prospective randomized trial. Eur J Gastroenterol Hepatol. 2021 Dec 1;33(1S Suppl 1):e909-e915. doi: 10.1097/MEG.0000000000002300. PMID 35048657